CLINICAL TRIAL: NCT02327208
Title: Effects of Carbohydrate and Protein Supplementation on Whole-body Protein Balance and Skeletal Muscle Mass During Winter Military Training: a Randomized Controlled Trial
Brief Title: Lean Body Mass Response to Higher-protein Diets During Winter Military Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stefan Pasiakos, Nutritional Physiologist, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-33HC
Record Dates: First submitted 2014-12-17; First posted 2014-12-30 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2015-04

CONDITIONS: Body Weight
Keywords: Military Training; Whey Protein; Body Composition
MeSH Terms: conditions — Body Weight | interventions — Proteins; Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): 3 Combat rations only per day. No additional experimental food items (those assigned to the active comparator groups will consume isoenergetic carbohydrate and protein-based food products).
  Interventions: Dietary Supplement: Control
- Protein (Active Comparator): Consume 4 whey protein-based snack-bars in addition to 3 combat rations each day during training.
  Interventions: Dietary Supplement: Protein
- Carbohydrate (Active Comparator): Consume 4 carbohydrate-based snack-bars in addition to 3 combat rations each day during training.
  Interventions: Dietary Supplement: Carbohydrate

INTERVENTIONS:
Dietary Supplement: Control
  Other Names: Placebo (Rations Only)
  Arms: Control
Dietary Supplement: Protein
  Other Names: Protein Bar
  Arms: Protein
Dietary Supplement: Carbohydrate
  Other Names: Granola Bar
  Arms: Carbohydrate

SUMMARY:
The objectives of this study are to: 1) determine effects of a prototype recovery food product providing supplemental energy on whole-body protein balance, skeletal muscle mass, and biomarkers of physiological status and strain during winter military training, and 2) determine the extent to which varying macronutrient composition (protein-based [PRO] versus carbohydrate-based [CHO]) of the food product modulates the physiological consequences to strenuous military training.

DETAILED DESCRIPTION:
Up to 120 Norwegian Soldiers from the 2nd Battalion, Brigade North, Norwegian Army stationed at Skjold Garrison will be enrolled in a 9-day, randomized controlled study. Using dietary analysis, body composition assessments, stable isotope methodologies, basic biochemical techniques, and measures of physiological strain, the effects of supplemental energy in the form of carbohydrate and protein on indices of muscle mass and physiological status will be assessed.

We hypothesize that consuming supplemental energy will attenuate the effects of severe energy deficit on inflammation, androgenic hormones, and whole-body protein retention, thereby protecting skeletal muscle mass. We expect that consuming PRO will promote a more favorable recovery than consuming CHO, as indicated by measures of increased whole-body protein synthesis and greater conservation of skeletal muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Norwegian Soldiers aged 18 years or older participating in the 4-day training program.

Exclusion Criteria:

* History of skin irritation (e.g., nickel or adhesive allergy), difficulty swallowing large pills, and allergies to dairy products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Protein Balance | day 5
  Whole-body nitrogen balance
Lean Body Mass | day 5
  Body composition
Skeletal Muscle Mass | day 5
  Isotopic estimates of muscle protein mass
Body weight | day 5

SECONDARY OUTCOMES:
Intestinal health | day 5
  Gut health
Thermal and Physiological Strain | average 6 days
  Core and skin temperature, heart rate, respiration rate

CONTACTS AND LOCATIONS:
Locations (3):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States
- Norway (2):
  - Norwegian Defense Research Establishment, Kjeller
  - Skjold Garrison, Skjold

REFERENCES:
- [Background] Karl JP, Margolis LM, Madslien EH, Murphy NE, Castellani JW, Gundersen Y, Hoke AV, Levangie MW, Kumar R, Chakraborty N, Gautam A, Hammamieh R, Martini S, Montain SJ, Pasiakos SM. Changes in intestinal microbiota composition and metabolism coincide with increased intestinal permeability in young adults under prolonged physiological stress. Am J Physiol Gastrointest Liver Physiol. 2017 Jun 1;312(6):G559-G571. doi: 10.1152/ajpgi.00066.2017. Epub 2017 Mar 23. PMID 28336545
- [Result] Margolis LM, Murphy NE, Martini S, Gundersen Y, Castellani JW, Karl JP, Carrigan CT, Teien HK, Madslien EH, Montain SJ, Pasiakos SM. Effects of Supplemental Energy on Protein Balance during 4-d Arctic Military Training. Med Sci Sports Exerc. 2016 Aug;48(8):1604-12. doi: 10.1249/MSS.0000000000000944. PMID 27054679
- [Result] Pasiakos SM, Margolis LM, Murphy NE, McClung HL, Martini S, Gundersen Y, Castellani JW, Karl JP, Teien HK, Madslien EH, Stenberg PH, Young AJ, Montain SJ, McClung JP. Effects of exercise mode, energy, and macronutrient interventions on inflammation during military training. Physiol Rep. 2016 Jun;4(11):e12820. doi: 10.14814/phy2.12820. PMID 27273884